CLINICAL TRIAL: NCT06260085
Title: The Effect of Listening to the Voice Recording of Relatives on Chest Pain, Anxiety and Depression in Patients Hospitalised in Coronary Intensive Care Unit: Randomised Controlled Study
Brief Title: Effect of Listening to Relatives' Voice Recordings on Chest Pain, Anxiety, and Depression in Coronary ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Yasemin Kalkan Uğurlu, Assist Prof., Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 686
Record Dates: First submitted 2024-01-25; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Acute Myocardial Infarction; Intensive Care Unit Syndrome
Keywords: Acute myocardial infarction; Anxiety; Chest pain; Voice recording
MeSH Terms: conditions — Anxiety Disorders; Chest Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The clinical nurse collected the data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): After the condition of the patients in the control group was stable, the pre-test was administered, then the patient was given routine information (Your mother/father/daughter/son/... is at the door, is there anything you want to tell them? I can convey and give feedback.). After the information, two more tests were administered at 15 and 30 minutes.
- İntervention (Experimental): In this randomised, controlled, experimental study, patients were randomised into intervention and control groups according to gender and age groups. In the preliminary interviews with the family members of the patients in the intervention group, the message content was discussed with the relatives of the patients before the voice recording was taken and carefully prepared to prevent negative effects. After the patient's condition was stable, the pretest was administered 15 minutes before (T1) the voice recording of the patient's relative was played through the music pillow.After the application, two more tests were applied at 15 (T2) and 30 (T3) minutes.
  Interventions: Other: Relatives vioce record

INTERVENTIONS:
Other: Relatives vioce record — In the study, it was emphasized that the messages to be played to the patient should be 3-5 minutes and simple terms should be used in a way that can be understood by individuals with low education level. Written informed consent was obtained from the patient and the patient's relatives before the application. In the message recorded by a patient's relative decided by the patient's family members, the patient's relative said what he/she wanted to say to the patient and recorded it using a voice recorder. The researcher had a preliminary interview with the patient's relative before the voice recording was taken about the use of the voice recorder and the content of the message (Table 1) in order to prevent the messages from negatively affecting the patient. The voice recording created by the patient's relative was played to the patient by the researcher using a music pillow. After the patient listened to the audio recording, it was erased under the witness of the patient's relative.
  Arms: İntervention

SUMMARY:
The aim of the study was to evaluate the effect of listening to the voice recordings of relatives of patients with acute myocardial infarction (AMI) who were treated in the coronary intensive care unit on chest pain, anxiety and depression parameters of the patients.

Methods In the study, which was conducted as a randomised, controlled, experimental study, voice recordings of the family members of the patients were created and played to the patients through a music pillow. The study was carried out with 60 patients, 30 experimental and 30 control groups. Three tests were applied to the patients 15 minutes before, 15 and 30 minutes after the application. The data of the study were collected using the "Patient Introduction Form", "Hospital Anxiety Depression Scale", "Visual Analogue Scale" and "Patient Follow-up Form".

DETAILED DESCRIPTION:
In the study, it was emphasized that the messages to be played to the patient should be 3-5 minutes and simple terms should be used in a way that can be understood by individuals with low education level. Written informed consent was obtained from the patient and the patient's relatives before the application. In the message recorded by a patient's relative decided by the patient's family members, the patient's relative said what he/she wanted to say to the patient and recorded it using a voice recorder. The researcher had a preliminary interview with the patient's relative before the voice recording was taken about the use of the voice recorder and the content of the message in order to prevent the messages from negatively affecting the patient. The voice recording created by the patient's relative was played to the patient by the researcher using a music pillow. After the patient listened to the audio recording, it was erased under the witness of the patient's relative.In this randomised, controlled, experimental study, patients were randomised into intervention and control groups according to gender and age groups. In the preliminary interviews with the family members of the patients in the intervention group, the message content was discussed with the relatives of the patients before the voice recording was taken and carefully prepared to prevent negative effects. After the patient's condition was stable, the pretest was administered 15 minutes before (T1) the voice recording of the patient's relative was played through the music pillow.After the application, two more tests were applied at 15 (T2) and 30 (T3) minutes. After the condition of the patients in the control group was stable, the pre-test was administered, then the patient was given routine information (Your mother/father/daughter/son/... is at the door, is there anything you want to tell them? I can convey and give feedback.). After the information, two more tests were administered at 15 and 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Adult age group (over 18 years),
* Not being diagnosed with psychiatric and neurological diseases,
* Diagnosis of AMI by a cardiologist,
* First time in the coronary intensive care unit,
* It's his first AMI,
* Being able to speak and understand Turkish.

Exclusion Criteria:

* Known hearing problems,
* Previous cardiovascular disease and history of myocardial infarction,
* Previous coronary artery bypass surgery and/or percutaneous transluminal coronary angioplasty to be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-04 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Chest Pain | 15 minutes before (T1), 15 minutes later (T2), 30 minutes later (T3)
  Patients' chest pain was assessed using a visual analog scale (VAS). The VAS consists of a 10 cm horizontal line ranging from 0 to 10, with zero indicating the lowest level of pain and 10 indicating the highest level. Patients were asked to describe the intensity of chest pain on a scale of 0-10. The VAS criterion is very effective, valid and reliable in determining the intensity of pain. The VAS is also a standardized scale for measuring anxiety with appropriate validity and reliability that has been used in various studies

SECONDARY OUTCOMES:
Anxiety, and Depression | 15 minutes before (T1), 15 minutes later (T2), 30 minutes later (T3)
  Patients' anxiety and depression was assessed using The Hospital Anxiety Depression (HAD) Scale was developed by Zigmond and Snaith (1983) to determine the patient's risk for anxiety and depression and to measure the level and severity change .As a result of the validity and reliability study, the cut-off score for the anxiety subscale (HAD-A) was 10 and the cut-off score for the depression subscale (HAD-D) was 7. Accordingly, those who score above these points are considered to be at risk. The scale is a four-point Likert-type scale and the total scale score is scored between 0-42.

CONTACTS AND LOCATIONS:
Locations (1):
- Yasemin Kalkan Uğurlu, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No